CLINICAL TRIAL: NCT01287377
Title: Smoking Cessation With the Nicotine Patch: A Pilot Study of Patch Messaging
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100683
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: tobacco cessation; smoking cessation; nicotine; counseling; telephone; self-help; smoking abstinence; tobacco use disorder; nicotine replacement therapy
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pre-Patch and Telephone Counseling (Experimental): Nicotine patches (2 weeks' worth) are mailed directly to the subject. Clients will be encouraged to start using these patches PRIOR to their quit date.
  Counseling includes a comprehensive pre-quit session (to include motivation, planning, discussion of nicotine patch use, and setting of a quit date) and up to 4 proactive follow-up calls.
  Interventions: Behavioral: Telephone Counseling; Drug: Nicotine Patches
- Post-Patch and Telephone Counseling (Active Comparator): Nicotine patches (2 weeks' worth) are mailed directly to the subject. Clients are encouraged to start using their patches ON their quit date.
  Counseling includes a comprehensive pre-quit session (to include motivation, planning, discussion of nicotine patch use, and setting of a quit date) and up to 4 proactive follow-up calls.
  Interventions: Behavioral: Telephone Counseling; Drug: Nicotine Patches
- Telephone Counseling and no patches sent (Active Comparator): Counseling includes a comprehensive pre-quit session (to include motivation, planning, discussion of nicotine patch use, and setting of a quit date) and up to 4 proactive follow-up calls.
  Interventions: Behavioral: Telephone Counseling

INTERVENTIONS:
Behavioral: Telephone Counseling — Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
Drug: Nicotine Patches — Subjects are randomized into one of these pharmacotherapy interventions: direct mailing of active patches with a message to start using it on their quit date, direct mailing of active patches with a message to start using it right away, or usual care patches in which no patches are sent directly (although clients may still get them through their usual channels).
  For those in the usual care condition, patches will not be mailed directly to them; however, we will facilitate their use by providing a certificate that can be used by the State Medicaid program and some other insurance companies to obtain free patches. For those in the active condition, we will mail 2 weeks of patches directly to their home. All subjects will receive a 2 week starter kit with fourteen 21mg patches.
  Other Names: Habitrol
  Arms: Post-Patch and Telephone Counseling; Pre-Patch and Telephone Counseling

SUMMARY:
The primary purpose of this study is to test the feasibility of sending pre-cessation nicotine patches and to examine the effects associated with the pre-cessation treatment phase. Specifically, this study aims to:

1. See if subjects will use pre-cessation nicotine patches.
2. See if subjects in the pre-cessation nicotine patches go on to get more nicotine patches.
3. See if pre-cessation treatment with nicotine patches leads to a decrease in number of cigarettes smoked per day.
4. See if sending 2-weeks' worth of patches is helpful to the quitting process.

DETAILED DESCRIPTION:
Quitlines have become central to state tobacco control efforts in the U.S. In addition to offering telephone counseling, many quitlines have begun providing quitting aids (e.g., nicotine patch) to eligible smokers. The nicotine patch has been shown repeatedly to double the rate of quitting success compared to a placebo control. Recently a number of studies have examined the use of patches prior to quitting. A meta-analysis indicates that such pre-cessation treatment with nicotine patches doubles the odds of quitting, compared to starting patch treatment on the quit day, as is traditionally done.

The proposed study would look at both pre-cessation treatment with nicotine patches as well as looking to see if sending clients nicotine patches is helpful in their quitting process. The rationale for pre-cessation treatment with patches is that using patches in this manner would make it easier to quit smoking because it may: reduce the reinforcing effects of cigarette smoking, thus helping to overcome conditioned behavior; reduce the need for inhaled nicotine as smokers naturally decrease their cigarette consumption to titrate the level of nicotine in their system; and/or increase compliance with patch use in the quitting phase.

The rationale for sending nicotine patches is that when callers must go and get the patches on their own it creates a barrier to their quitting so that sending nicotine patches directly to a callers' home would make it easier for them to stay on task and quit. This pilot will allow us to test the feasibility of sending pre-treatment nicotine patches and to examine the effects associated with the pre-cessation treatment phase.

This pilot project has the following specific aims, to examine whether:

1. Subjects will use pre-cessation nicotine patches.
2. Subjects in the pre-cessation nicotine patches go on to get more nicotine patches.
3. Pre-cessation treatment with nicotine patches leads to a decrease in number of cigarettes smoked per day.
4. Sending 2-weeks' worth of patches is helpful to the quitting process.

Results will add to the theoretical understanding of behavior change from which new, effective interventions can spring.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years old
* Daily smoker
* >=10 cigarettes per day
* Ready to quit within one month
* First time quitline caller
* Valid phone number
* Valid address (no P.O. boxes)
* California resident
* Agree to participate in study and evaluation
* English speaking

Exclusion Criteria:

* Uses other form of tobacco
* Plan to use quitting aids other than nicotine patch
* Has any of the following conditions:
* Severe allergy to adhesive tape
* Arrhythmia
* Angina
* Heart attack within last 6 months
* Stroke within last 6 months
* Uncontrolled high blood pressure
* Insulin-dependent diabetes
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — UCSD
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from 11/8/2010 - 1/18/2011
Groups:
- Pre-Patch and Telephone Counseling: 2-weeks of nicotine patches mailed directly to the subject. Clients will be encouraged to start using these patches PRIOR to their quit date.
  Counseling includes a comprehensive pre-quit session (to include motivation, planning, discussion of nicotine patch use, and setting of a quit date) and up to 4 proactive follow-up calls.
  Telephone Counseling: Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
  Nicotine Patches: Subjects are randomized into one of these pharmacotherapy interventions: direct mailing of active patches with a message to start using it on their quit date, direct mailing of active patches with a message to st
- Post-Patch and Telephone Counseling: 2-weeks of nicotine patches mailed directly to the subject. Clients are encouraged to start using their patches ON their quit date.
  Counseling includes a comprehensive pre-quit session (to include motivation, planning, discussion of nicotine patch use, and setting of a quit date) and up to 4 proactive follow-up calls.
  Telephone Counseling: Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
  Nicotine Patches: Subjects are randomized into one of these pharmacotherapy interventions: direct mailing of active patches with a message to start using it on their quit date, direct mailing of active patches with a message to start usi
Period: Overall Study
Arm/Group | Pre-Patch and Telephone Counseling | Post-Patch and Telephone Counseling | Telephone Counseling and no Patches Sent
Started | 80 | 81 | 82
Completed | 80 (Study Complete) | 81 (Study Complete) | 82 (Study Complete)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-Patch and Telephone Counseling: Nicotine patches (2 weeks' worth) are mailed directly to the subject. Clients will be encouraged to start using these patches PRIOR to their quit date.
  Counseling includes a comprehensive pre-quit session and up to 4 proactive follow-up calls.
  Telephone Counseling: Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
- Post-Patch and Telephone Counseling: Nicotine patches (2 weeks' worth) are mailed directly to the subject. Clients are encouraged to start using their patches ON their quit date.
  Counseling includes a comprehensive pre-quit session and up to 4 proactive follow-up calls.
  Telephone Counseling: Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
- Telephone Counseling and no Patches Sent: Counseling includes a comprehensive pre-quit session and up to 4 proactive follow-up calls.
  Telephone Counseling: Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
  Patches will not be mailed directly to them; however, we will facilitate their use by providing a certificate that can be used by the State Medicaid program and some other insurance companies to obtain free patches.
- Total: Total of all reporting groups
Arm/Group | Pre-Patch and Telephone Counseling | Post-Patch and Telephone Counseling | Telephone Counseling and no Patches Sent | Total
Number analyzed (Participants) | 80 | 81 | 82 | 243
Age, Customized [Count of Participants; unit: Participants]
  18-24 | 7 | 9 | 7 | 23
  25-44 | 35 | 30 | 39 | 104
  45-64 | 35 | 40 | 33 | 108
  65+ | 3 | 2 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 52 | 143
  Male | 34 | 36 | 30 | 100
Education >12 Year [Count of Participants; unit: Participants] | 42 | 36 | 44 | 122

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have Not Used Tobacco in the Past 30 Days
Description: At a given point in time (in this case, 2 months after program registration), quitline participants are asked whether they have used cigarettes or other forms of tobacco in the past 30 days. Those who reply that they have not used tobacco in the past 30 days are considered to have quit.
Time Frame: 2-months post enrollment
Population: The number of participants analyzed is the number of participants the quitline was able to reach at 2-months post enrollment, not the number randomized into that condition
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Patch and Telephone Counseling | Post-Patch and Telephone Counseling | Telephone Counseling and no Patches Sent
Number analyzed (Participants) | 60 | 65 | 60
Participants | 18 | 26 | 10

2. Secondary Outcome: Number of Participants With Serious Quit Attempts
Description: A serious quit attempt is considered is a quit attempt that last more than 24 hours
Time Frame: 2-months post enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Patch and Telephone Counseling | Post-Patch and Telephone Counseling | Telephone Counseling and no Patches Sent
Number analyzed (Participants) | 60 | 65 | 60
Participants | 48 | 53 | 42

ADVERSE EVENTS:
Groups:
- Pre-Patch and Telephone Counseling: Nicotine patches (2 weeks' worth) are mailed directly to the subject. Clients will be encouraged to start using these patches PRIOR to their quit date.
  Counseling includes a comprehensive pre-quit session (to include motivation, planning, discussion of nicotine patch use, and setting of a quit date) and up to 4 proactive follow-up calls.
  Telephone Counseling: Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
  s.
- Post-Patch and Telephone Counseling: Nicotine patches (2 weeks' worth) are mailed directly to the subject. Clients are encouraged to start using their patches ON their quit date.
  Counseling includes a comprehensive pre-quit session (to include motivation, planning, discussion of nicotine patch use, and setting of a quit date) and up to 4 proactive follow-up calls.
  Telephone Counseling: Telephone counseling has several distinguishing features, namely proactive follow up counseling calls, a manualized protocol, and relapse-sensitive scheduling. The follow-up call schedule includes a reminder call if the quit date is more than one week out, a call within 24 hours of the quit attempt, another call 4-7 days after the quit date, and another call 10-14 days after the quit date.
Arm/Group | Pre-Patch and Telephone Counseling | Post-Patch and Telephone Counseling | Telephone Counseling and no Patches Sent
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/81 | 0/82
Other Adverse Events (participants affected / at risk) | 0/80 | 0/81 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No